CLINICAL TRIAL: NCT03621007
Title: An Observational,Prospective Natural History Study of Early-Onset Extreme Obesity Due to Bi-Allelic Loss-of-Function Mutations in the POMC, PCSK1 or LEPR Genes
Acronym: NHS
Status: Completed | Type: Observational
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RM-493-016
Record Dates: First submitted 2018-07-30; First posted 2018-08-08 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: POMC Deficiency Obesity; PCSK1 Deficiency Obesity; LEPR Deficiency Obesity
Keywords: POMC; LEPR; PCSK1; Bi-Allelic Loss; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- POMC deficiency obesity
- LEPR deficiency obesity
- PCSK1 deficiency obesity

SUMMARY:
This is an observational study. There are no protocol-defined visits, although patients are expected to have routine office visits approximately every 6 months. Upon signing of informed consent/assent and study enrollment, historical data will be abstracted from the patient's medical chart. The patient will then be observed prospectively for up to 5 years, with additional data collected from routine healthcare encounters and direct-to-patient questionnaires (where local laws allow), including laboratory tests, physical exam and patient reported outcomes/quality of life measures. Patients will be consented/assented to provide blood samples for biomarker assessments, DNA sequencing and archiving.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 years or older
2. Study participant and/or parent or guardian is able to communicate well with the investigator, to understand and comply with the requirements of the study, and be able to understand and sign the written informed consent/assent.
3. Have documented results of DNA sequencing for the three genes of interest: POMC, PCSK1 and LEPR.
4. Bi-allelic, homozygous or compound heterozygous (a different gene mutation on each allele) genetic status for either the POMC or PCSK1 genes, resulting in a severe POMC deficiency obesity clinical phenotype, or a similar bi-allelic gene status for the LEPR gene leading to identified LEPR deficiency obesity.
5. Patients who are willing to come in for routine office visits approximately every 6 months.

Exclusion Criteria:

1. Participation within the past 3 months in a clinical trial of any investigational medicine for obesity.
2. Confirmed diagnosis of Prader-Willi syndrome, Bardet-Biedl syndrome, Alström syndrome, or other syndromic form of genetic obesity.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with POMC, PCSK1 or LEPR deficiency obesity due to a bi-allelic loss of function genetic mutation will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Demographics | Baseline
  Descriptive summary of baseline characteristics including age, sex, ethnicity, and race.
Medical history | 5 years
  Descriptive summary of medical history over time.
Clinical course | 5 years
  Descriptive summary of disease progression over time.

CONTACTS AND LOCATIONS:
Overall Officials: Murray Stewart, MD, Study Chair — Rhythm Pharmceuticals, Inc
Locations (3):
- Turkey (Türkiye) (3):
  - Dokuz Eylul Universitesi Tip Fakultesi, Balçova
  - Ege University School of Medicine of Pediatric Endocrinology, Bornova
  - Pediatric Endocrinology and Diabetes Marmara University Hospital, Istanbul